CLINICAL TRIAL: NCT04019847
Title: A Feasibility Study Considering the Use of the STAK Tool in Addition to Standard Physiotherapy Compared to Standard Physiotherapy Alone to Treat Arthrofibrosis Patients Following Total Knee Replacement
Brief Title: STAK Tool for Treatment of Arthrofibrosis Post Total Knee Replacement
Acronym: STAK
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospitals, Leicester (Other)
Responsible Party: Principal Investigator, Sara Aspinall, Principal Investigator, University Hospitals, Leicester
Allocation: Non-Randomized | Model: Sequential | Masking: Single | Purpose: Treatment
Other Study IDs: 93160
Record Dates: First submitted 2018-06-11; First posted 2019-07-15 (Actual); Last update posted 2020-04-28 (Actual); Status verified 2020-04

CONDITIONS: Arthrofibrosis

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- STAK Tool (Experimental): The STAK Tool enables patients to apply a high intensity stretch to their knee independently. Patients are asked to do this for a maximum of 60 mins per day.
  Interventions: Device: STAK Tool; Other: Standard treatment
- Standard treatment (Active Comparator): Patients are treated as per their Clinician's prescription. Physiotherapists tailor treatment of arthrofibrosis to meet their patients' individual needs. Treatment may comprise the following: education, advice and a range of stretching exercises/techniques to change the length and density of the adhesions and shortened tissue. These include active range of movement (AROM), passive range of movement (PROM), strengthening exercises, hands-on high intensity passive physiological stretches, joint mobilisations and a home exercise programme involving full weight bearing exercises with the aim of enabling the patient to regain ROM and function.
  Interventions: Other: Standard treatment

INTERVENTIONS:
Device: STAK Tool — Medical stretching device
  Arms: STAK Tool
Other: Standard treatment — Physiotherapists tailor treatment of arthrofibrosis to meet their patients' individual needs. Treatment may comprise the following: education, advice and a range of stretching exercises/techniques to change the length and density of the adhesions and shortened tissue. These include active range of movement (AROM), passive range of movement (PROM), strengthening exercises, hands-on high intensity passive physiological stretches, joint mobilisations and a home exercise programme involving full weight bearing exercises with the aim of enabling the patient to regain AROM and function

SUMMARY:
A common complication following total knee replacement (TKR) is arthrofibrosis, a severe stiffening of the knee caused by scar tissue.

The aims of this mixed methods feasibility study are to (1) record the effect of use of the STAK Tool on knee flexion active range of movement (KROM) immediately following 8 weeks use and 6 months following use, (2) explore patients' experiences of arthrofibrosis and use of the STAK Tool, (3) Consider appropriate outcome measures (e.g. KROM, patient experience/acceptability, The Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC), Oxford Knee Score (OKS) and other clinical measures and (4) design a protocol to evaluate the effectiveness of the STAK Tool.

DETAILED DESCRIPTION:
Arthrofibrosis most commonly occurs after total knee replacement (TKR), extensive intra-articular injury or surgical procedures, for example fracture of the proximal tibia or distal femur or multiple ligament reconstructions (Creighton and Bach 2012). Arthrofibrosis involves a severe stiffening of the knee caused by scar tissue. This often results in a lack of crucial range of knee flexion movement. Traditional physiotherapy treatment includes a home exercise programme involving regular intense stretches and mobilisations delivered by the physiotherapist at the hospital aiming to enable the patient to regain optimal, functional knee bend. The inflammatory process and remodeling of soft tissues following trauma can lead to production of scar tissue and subsequent stiffness. This results in increased pain and difficulty in performing exercises. This often limits progress requiring high numbers of physiotherapy sessions and potentially further surgery (manipulation under anaesthetic) to restore range of movement.

The STAK Tool enables the patient to perform intense self-stretching of the knee more easily and effectively. Intense stretching is essential to increase KROM (Bonutti et al 2008, Bonutti 2010, Papotto et al 2012, Stephenson et al 2010). Patients who fall into the category of having restricted KROM (less than 70 degrees flexion) and those whose Clinicians identify them as requiring further intensive physiotherapy to address their stiffness would be approached to take part in this study. 36 participants would be recruited. Participants would be over 18 years old, between 44kg and 159kg. This mixed methods feasibility study would investigate patients' progress and outcomes in overcoming arthrofibrosis using the STAK Tool a medical stretching device at home plus standard physiotherapy treatment (intervention group), compared to patients receiving physiotherapy treatment only (comparative group). Participants would be allocated into either the intervention or comparative group. Participants would be instructed to use the STAK Tool for 5-10 minute periods for a minimum total of 20 minutes and maximum of 60 minutes a day.

Participants would receive their standard physiotherapy treatment including KROM, full weight bearing exercises including sit to stands, squats, body weight assisted passive stretches, strengthening exercises and mobilisations. Angle of knee flexion would be measured (standardised method) by the Principal Investigator and the WOMAC and OKS are administered on the day the participant consents to the study (Visit 1), the day the intervention starts. This will be within approximately 2 weeks of the patient being identified by their clinician. (The Principal investigator will visit the participant within 10 days to ensure there are no problems using the STAK Tool (Visit 2 - only intervention group). During Visit 1 an interview (interview 1), would be conducted to explore the patients' initial thoughts on the STAK Tool after being introduced to it. Both the intervention and comparative groups will have their KROM recorded using two different measuring instruments, the universal goniometer and the Hudl Ubersense App. Outcome measures including KROM, WOMAC and OKS will be recorded again following approximately 8 weeks treatment (dependent on time available before manipulation as per normal clinical care), at either the patient's final follow-up with their Clinician or at their home (Visit 3) (end of intervention). The WOMAC and OKS would help to ascertain the patient's perceptions of pain, stiffness and functional improvements. At Visit 3 participants would also complete a questionnaire regarding the frequency of knee stretching exercise completed and how easy/difficult it had been to achieve. On completing 8 weeks standard treatment patients in the comparative group who were deemed eligibility by their Clinician would be offered the STAK Tool 8 week treatment.

Visits would then be completed as per the intervention group minus the interviews.

An in-depth semi-structured interview (interview 2) will be conducted with participants in the intervention group exploring their thoughts and experiences of using the STAK Tool to increase their knee flexion, their perceived progress and acceptability of the device.

A follow up meeting (Visit 4) would take place at 6 months after Visit 3, this would take place at the participant's home patients KROM, WOMAC and OKS would be recorded to provide data relating to participants long term outcomes.

ELIGIBILITY:
Inclusion Criteria:

* male or female,
* 18 to 95 year olds,
* having received a primary total knee replacement within the last 12 months.
* Following their TKR have less than 70 degrees knee flexion or have been prescribed intensive physiotherapy for their knee stiffness by their Consultant.
* Between 44kg and 159kg.

Exclusion Criteria:

* post malignancy or knee trauma
* have leaking wounds or infected joints,
* have rheumatoid arthritis or osteoporosis,
* have undergone long term steroid treatment or the clinician felt the patient was at risk of post-operative fracture.
* Fell outside weight limits (44kg to 159kg),
* Unable to give consent themselves (confusion, non-English speaking patients).

Ages: 18 Years to 95 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2017-08-02 (Actual); Primary Completion 2019-08-19 (Actual); Study Completion 2019-08-19 (Actual)

PRIMARY OUTCOMES:
Change in range of knee movement as assessed using a universal goniometer | Baseline, 8 weeks after intervention/control, and 6 months after intervention/control
  Universal goniometer used to measure knee range of movement
Change in range of knee movement as assessed using a mobile app. | Baseline, 8 weeks after intervention/control, and 6 months after intervention/control
  A Mobile app used to measure knee range of movement

SECONDARY OUTCOMES:
WOMAC Score (The Western Ontario and McMaster Universities Osteoarthritis Index) | Baseline, 8 weeks after intervention/control, and 6 months after intervention/control
  Patient reported outcome measure relating to patient's pain, stiffness and function
Oxford Knee Score (OKS) | Baseline, 8 weeks after intervention/control, and 6 months after intervention/control
  Patient reported outcome measure relating to pain and function, specifically designed for total knee replacement patients.

OTHER OUTCOMES:
Semi-structured interviews | Prior to and following use of the STAK Tool for 8 weeks
  Two Semi-structured interviews conducted with intervention group to understand their experiences of having arthrofibrosis and their thoughts on the STAK Tool treatment.
Home exercise questionnaire | Immediately following intervention period.
  Questionnaire to capture patient's adherence to treatment, what this has involved, record changes in pain relief.
  This is a bespoke questionnaire designed by the researchers. It does not have a scale producing a final score. It provides additional information about adherence and intensity of exercise which will help us to better understand the reason for changes in range of movement
Acceptability Questionnaire | Immediately following STAK Tool intervention period.
  Questionnaire regarding acceptability of the STAK Tool to patients. Questionnaire to capture patient's adherence to treatment, what this has involved, record changes in pain relief.
  This is a bespoke questionnaire designed by the researchers. It does not have a scale producing a final score.

CONTACTS AND LOCATIONS:
Overall Officials: Sara Aspinall, MScR, Principal Investigator — University Hospitals, Leicester
Locations (1):
- University Hospitals of Leicester NHS Trust, Leicester, United Kingdom